CLINICAL TRIAL: NCT01184963
Title: Effect of High-protein or Normal-protein Diet on Weight Loss, Body Composition, Hormone and Metabolic Profile in Women With Polycystic Ovary Syndrome From South Brazil: A Randomized Study
Brief Title: High Versus Normal Protein Diet in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Poli Mara Spritzer, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-364
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2009-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; High protein diet
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controls (Other): Women in reproductive age regular ovulatory cycles
  Interventions: Dietary Supplement: High protein diet; Dietary Supplement: Normal protein diet
- PCOS patients (Other): Patients with anovulatory cycles, hyperandrogenism with or without polycystic ovarian appearance
  Interventions: Dietary Supplement: High protein diet; Dietary Supplement: Normal protein diet

INTERVENTIONS:
Dietary Supplement: High protein diet — High protein diet (30% protein, 40% carbohydrate, 30% lipid)
Dietary Supplement: Normal protein diet — Normal protein diet (15% protein, 55% carbohydrate, 30% lipid

SUMMARY:
The objective of this study is to assess the effects of a high protein (HP) and a normal protein diet (NP) on patients with polycystic ovary syndrome (PCOS) and body mass index (BMI)-matched controls in a sample of southern Brazilian women.

Patients will be randomized to receive high protein (30% protein, 40% carbohydrate, 30% lipid) or normal protein (15% protein, 55% carbohydrate, 30% lipid) during eight weeks.

The investigators hypothesis is that a different diet composition may have influences in changes of the main characteristics of PCOS, like hyperandrogenism and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* women of reproductive age
* BMI ranging from 18.5 to 39.9 kg/m²

Exclusion Criteria:

* Use of any drugs known to interfere with hormone levels for at least 3 months before the study
* Women with known type 2 diabetes, liver or renal disease or thyroid dysfunction
* Other hyperandrogenic disorders than PCOS

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in corporal weight | 8 weeks

SECONDARY OUTCOMES:
Changes in body composition | 8 weeks
changes in hormone and metabolic profile. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Poli Mara Spritzer, PhD, MD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil